CLINICAL TRIAL: NCT05064462
Title: Association Between TTV Viral Load and the Occurrence of Infections and Rejection in Heart Transplant Recipients
Brief Title: TTV Viral Load in Heart Transplant Recipients
Acronym: TTVCoeur
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: BioMérieux (Industry)
Responsible Party: Sponsor
Other Study IDs: APHP201167; 2020-A03456-33 (Other: IDRCB)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Heart Transplant Rejection; Heart Transplant Infection; Virus
Keywords: TTV, Heart transplant, Viral Load, rejection, infection
MeSH Terms: conditions — Virus Diseases; Langer-Giedion Syndrome; Rejection, Psychology; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5-7 ml whole blood samples are taken at each monthly visit to measure viral load at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All the patients included in the study: 50 patients, at least 18 years old, first heart transplant
  Interventions: Other: Collection of EDTA blood sample (5 to 7 ml)

INTERVENTIONS:
Other: Collection of EDTA blood sample (5 to 7 ml) — For all the patients included in the study, the samples to measure the viral load will be taken during the transplantation, then at each of the consultations planned as part of the usual care during the first year post-transplant (at minimum once and maximum twice a month).
  These samples will be taken at the same time as those taken as part of standard care.

SUMMARY:
This prospective, multicenter, non-interventional trial aims to study the association between TTV viral load and the occurrence of rejection or infection during the first year after transplantation.

The TTV viral loads, taken once a month during the first year after the transplant, will be measured at the end of the study.

DETAILED DESCRIPTION:
TTV (Torque Teno Virus) is a ubiquitous virus that is not associated with any disease. A correlation exists between the level of TTV replication and the subject's immunocompetence: weak or non-existent in immunocompetents, very high in immunocompromised patients. In heart transplant patients, pharmacological dosing of immunosuppressants prevents their toxic manifestations but is not correlated with individual immune competence. Only clinical manifestations of overdose (infections) or under dosage (rejections) currently allow optimization of immunosuppressants. A predictive biomarker of these clinical manifestations upstream of their appearance would revolutionize the management of these patients.

The TTV fulfills the conditions to be an ideal biomarker: classic blood sampling, possible follow-up in all patients, low cost, carrying out the analysis on already existing molecular biology platforms, reproducibility of inter- and intra-laboratory results, defined thresholds for the reliable interpretation of the results.

We believe that this marker will provide the clinician with a useful tool for the management of immunosuppressants and the patient with personalized medicine which will allow their management to be individualized. If this study confirms the expected results, then it will allow, secondly, the setting up of interventional studies to validate the TTV viral load as a biomarker, and a tool for piloting immunosuppressive treatment.

The TTV viral load of heart transplant patients will be follow during the first year after transplantation.

A tube of blood will be taken during the transplant and then once or twice a month.

Samples will be taken at the same time as those taken as part of standard care. The TTV viral load will be measured at the end of the study.

The occurrence of events of interest (infections and rejections) will be collected at each corresponding visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Heart transplant only
* First transplant
* Patient not having objected to carrying out the research
* Affiliated to a French Health Insurance system.

Exclusion Criteria:

* Patient transplanted from more than one solid organ
* Patient who has already been transplanted before
* Patient under guardianship or curatorship
* Patient under legal protection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with first heart transplant
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-03-03 (Estimated); Study Completion 2024-03-03 (Estimated)

PRIMARY OUTCOMES:
Composite outcome : Infections or Rejections | 12 months
  The primary endpoint is a composite endpoint defined as time to infections (first and recurrences) or rejections (first and recurrences) within the 12 months post-transplant:
  * Infections are defined as viral Infections , bacterial and parasitic infections requiring the establishment of anti-infectious treatment or hospitalization
  * Rejections are defined as acute type 2R or 3R cell rejections according to the ISHLT classification

SECONDARY OUTCOMES:
TTV viral load | 3 months
  Monthly mean of TTV viral concentration load measured by quantitative PCR within 3 months
TTV viral load | 12 months
  Monthly mean of TTV viral concentration measured by quantitative PCR within 12 months
Infections | 12 months
  Time to viral infections , bacterial and parasitic infections requiring the establishment of anti-infectious treatment or hospitalization during the 12 months post-transplant.
Rejections | 12 months
  Time to rejections within the 12 months post-transplant defined as acute type 2R or 3R cell rejections according to the ISHLT classification.
Immunosuppressant level | 3 months
  Immunosuppressant pharmacological dosing
Immunosuppressant level | 12 months
  Immunosuppressant pharmacological dosing

CONTACTS AND LOCATIONS:
Overall Officials: Hélène PERE, Pharm D, PhD, Principal Investigator — Hôpital Européen Georges-Pompidou; David VEYER, Pharm D, PhD, Study Director — Hôpital Européen Georges-Pompidou
Locations (3):
- France (3):
  - Hôpital européen Georges Pompidou, Paris
  - CHU de Rennes, Rennes
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI based on a scientific project and scientific involvement of the PI team. Collaboration will be fostered. Data sharing must respect the agreements made with funders. Teams wishing obtain IPD must meet the sponsor and IP team to present scientific (and commercial) purpose, IPD needed, format of data transmission, and timeframe. Technical feasibility and financial support will be discussed before mandatory contractual agreement. Processing of shared data must comply with European General Data Protection Regulation (GDPR).